CLINICAL TRIAL: NCT06866990
Title: Exploratory Clinical Study on the Efficacy and Safety of Lactobacillus Johnsonii in the Treatment of Patients with Premature Ovarian Insufficiency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-1343
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — CbsT2 protein, Lactobacillus johnsonii

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus johnsonii (Experimental): Participants receive Lactobacillus johnsonii
  Interventions: Dietary Supplement: Lactobacillus johnsonii
- Placebo (Placebo Comparator): Participants receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus johnsonii — The investigational product is a probiotic containing Lactobacillus johnsonii. It is recommended to be stored under refrigerated conditions at approximately 4°C. Participants are instructed to take one sachet twice daily, dissolved in warm water, with a total daily oral dose exceeding 1×10¹¹ colony-forming units (CFU).
  Arms: Lactobacillus johnsonii
Other: Placebo — The placebo product contains the same excipients as the investigational product, except for the absence of Lactobacillus johnsonii. It is identical to the investigational product in appearance, color, weight, and taste. It is recommended to be stored under refrigerated conditions at approximately 4°C. The administration method is the same as that of the experimental group.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to explore the effectiveness and safety of Lactobacillus johnsonii in improving ovarian function and perimenopausal symptoms in patients with premature ovarian insufficiency (POI). The main questions it aims to answer are: ① To explore the effectiveness and safety of Lactobacillus johnsonii in improving ovarian function and perimenopausal symptoms in patients with POI; ② To explore the potential mechanism of action of Lactobacillus johnsonii in improving ovarian function and perimenopausal symptoms in patients with POI. Participants who meet all the inclusion criteria will be enrolled in the study and randomly assigned in a 1:1 ratio to either the Lactobacillus johnsonii group or the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 39 years;
2. Irregular menstruation or amenorrhea for > 4 months;
3. At least two serum baseline follicle-stimulating hormone (FSH) levels > 25 IU/L (with an interval of more than 4 weeks between measurements);
4. Willing to voluntarily participate in this study, sign the informed consent form, and comply with the investigation and follow-up;
5. Not having participated in other clinical trials within the past 3 months.

Exclusion Criteria:

1. Use of antibiotics or probiotics, prebiotics, and live bacterial preparations within the past month or during the intervention period;
2. Received hormone replacement therapy within the past 2 months;
3. Chromosomal abnormalities and genetic defects;
4. Iatrogenic premature ovarian insufficiency;
5. Stage IV endometriosis;
6. Uncontrolled endocrine diseases or autoimmune diseases;
7. Organic gastrointestinal diseases;
8. Infectious diseases of the reproductive, urinary, or digestive systems;
9. Severe cardiovascular, respiratory, renal, hematologic, endocrine, neurological, psychiatric, or other systemic diseases that the investigator believes may interfere with the study evaluation;
10. History of venous thromboembolism;
11. Allergic or intolerant to the components of the investigational probiotic product;
12. Allergic to two or more types of food/medications;
13. Refusal to provide written informed consent;
14. Other conditions deemed unsuitable for participation in the study by the investigator.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Ovarian function markers | 6 months
  Changes in sex hormone levels (including follicle-stimulating hormone, luteinizing hormone, estradiol, progesterone, testosterone, prolactin and anti-Müllerian hormone) and menstruation resumption.

SECONDARY OUTCOMES:
Changes in antral follicle counts | 6 months
Changes in perimenopausal symptom | 6 months
  MENQOL Score (Menopause-Specific Quality of Life Questionnaire)
Changes in mental and psychological status | 6 months
  DASS-21 Scale (Depression, Anxiety, and Stress Scale-21)
Achievement of pregnancy | 8 months
  Pregnancy outcomes achieved through natural or assisted conception methods include biochemical pregnancy, clinical pregnancy, miscarriage, and ectopic pregnancy.
Changes in the gut microbiota. | 6 months

IPD SHARING:
Plan to Share IPD: No